CLINICAL TRIAL: NCT04494659
Title: A Single Center, Single Arm, Open and Fixed Sequence Study to Investigate the Pharmacokinetic Effects of Rifampicin on Famitinib in Healthy Male Subjects
Brief Title: A Drug-drug Interaction Trial to Evaluate the Pharmacokinetics Effect of Rifampicin on Famitinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FMTN-I-105
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-07

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — famitinib; Rifampin

STUDY DESIGN:
Intervention Model Description: Repeated oral doses of Rifampicin on the pharmacokinetic profile of a single dose of Famitinib.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): single dose of Famitinib on Day 1, and co-administered with Rifampicin on Day 16
  Interventions: Drug: Famitinib capsule; Drug: Rifampicin capsule

INTERVENTIONS:
Drug: Famitinib capsule — single dose and co-administrated with Rifampicin capsule
  Other Names: SHR1020
Drug: Rifampicin capsule — repeated doses of Rifampicin capsule
  Other Names: Rifampicin

SUMMARY:
The primary objective of the study was to assess the effect of repeated oral doses of Rifampicin on the pharmacokinetic profile of a single dose of Famitinib.

The secondary objective of the study was to assess the safety of Famitinib given alone versus Famitinib co-administered with Rifampicin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged 18 to 50 years old at the date of signing the informed consent;
2. Male body weight ≥ 50kg, body mass index (BMI) within the range of 19 ~ 28 kg/m2 (including 19 and 28) (BMI= weight (kg)/height 2 (m2));
3. Subjects have no childbirth plans and agree to take effective contraceptive measures within 3 months of the last medication;
4. The subject can communicate well with the researcher, understand and comply with the requirements of the study, understand and sign the informed consent.

Exclusion Criteria:

1. History of or currently suffering from any serious clinical diseases such as diseases in circulatory system, endocrine system, nervous system, digestive system, respiratory system, genitourinary system, hematology, immunology, psychiatry, and metabolic abnormalities, or any other diseases may interfere with the test results;
2. Any surgery within 6 months before screening, or plan to perform surgery during the study period, or who have previously undergone any surgery that affects gastrointestinal absorption (including gastrectomy, bowel resection, gastric reduction surgery, etc.)
3. Blood donation or massive blood loss (≥200 mL), or received blood transfusion, or used blood products within 3 months before screening;
4. History of allergy to drugs, food or other substances;
5. Frequent use of sedatives, sleeping pills or other addictive drugs; History of drug abuse within 1 year prior to screening; Positive for urine drug abuse screening test;
6. Participated in any clinical trial and took the study drug within 3 months prior to the first administration;
7. Used any prescription drug or herbal tonic within 1 month before the first administration; Have used any over-the-counter (OTC) medicines, food supplements (including vitamins, calcium tablets, etc.) within 2 weeks prior to the first administration;
8. Those who had smoked more than 5 cigarettes per day in the previous 3 months before screening and could not stop using any tobacco products during the study period; Nicotinic test positive;
9. Frequent drinkers in the previous 6 months before screening, i.e., those who drink more than 14 units of alcohol per week (1 unit = 285 mL beer, or 25 mL spirits, or 100 mL wine) and cannot stop using any alcoholic products during the study period; alcohol test positive;
10. Abnormal vital signs, physical examination, 12-lead ECG, abdominal B-ultrasound, chest radiograph, routine blood test, biochemical test, routine urine test and blood coagulation test with clinical significance;
11. Hepatitis B surface antigen positive, hepatitis C antibody positive, syphilis antibody positive, HIV antibody positive;
12. Subjects have taken and do not agree to stop using any drink or food containing methylxanthine, such as coffee, tea, cola, chocolate, etc. from 48 hours before the first administration until end of the study;, subjects have taken and do not agree to discontinue any beverage or food containing grapefruit from 7 days prior to initial administration until end of the study; Those who have special requirements on diet and cannot follow a uniform diet;
13. Subjects who are considered to have other factors that are not appropriate to participate in this study by the investigator.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Cmax of Famitinib | Day 1 to Day 24
  Pharmacokinetics parameters of Famitinib
AUC0-t of Famitinib | Day 1 to Day 24
  Pharmacokinetics parameters of Famitinib
AUCinf of Famitinib | Day 1 to Day 24
  Pharmacokinetics parameters of Famitinib

SECONDARY OUTCOMES:
Tmax of Famitinib | Day 1 to Day 24
  Pharmacokinetics parameters of Famitinib
T1/2 of Famitinib | Day 1 to Day 24
  Pharmacokinetics parameters of Famitinib
CL/F of Famitinib | Day 1 to Day 24
  Pharmacokinetics parameters of Famitinib
Vz/F of Famitinib | Day 1 to Day 24
  Pharmacokinetics parameters of Famitinib
incidence of adverse events/serious adverse events | from ICF signing date to approximate Day 31
  safety evaluation based on NCI-CTC AE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li T, Li X, Jiang X, Wang C, Sun F, Liu Y, Lin P, Shi P, Fu Y, Gao X, Zhang Y, Cao Y. The effect of rifampin on the pharmacokinetics of famitinib in healthy subjects. Cancer Chemother Pharmacol. 2022 Nov;90(5):409-415. doi: 10.1007/s00280-022-04474-8. Epub 2022 Sep 15. PMID 36107220